CLINICAL TRIAL: NCT03721887
Title: Exploit the Neural Source and the Feasibility of Transcranial Direct Current Stimulation for Freezing of Gait in Parkinson's Disease and Multiple System Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The chief, Department of Neurology, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH106-REC2-171
Record Dates: First submitted 2018-09-17; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease; Multiple System Atrophy
Keywords: Parkinson's disease; Multiple system atrophy; Freezing of gait; Transcranial direct current stimulation
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): In transcranial direct current stimulation, the anodal pad was tapped over the primary motor cortex and the cathode pad was adhered of the contralateral frontal region. A constant current of 2.0 mA will be apply for up to 20 mins.
  Interventions: Device: Transcranial direct current stimulation
- sham tDCS (Sham Comparator): In transcranial direct current stimulation, the sham stimulation will be 30s stimulation with ramp up and ramp off for 10s at 2.0 mA.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — A consecutive 5-days course of tDCS will be delivered. In treatment group, true stimulation will be administrated and sham stimulation will be delivered in control group.

SUMMARY:
In this project, the investigators will deliver a 5-day session of transcranial direct current stimulation (tDCS) to the leg motor cortex of the FOG patients to examine whether the intervention will benefit the patients in a double blind randomized design. Six assessments with different combinations of clinical scaling, gait analysis, electrophysiological investigation and fMRI examinations before and after tDCS will be conducted. The treatment and placebo groups will be crossed over after one-month washout. The investigators will investigate whether the possible tDCS beneficial effect will be different or similar in patients with different electric sources. In addition, how long the possible beneficial effect of tDCS can be consolidated after the 5-day course of stimulation is also crucial. The investigators aim to peep the myth of FOG in PD and MSA by the multi-modality approach and hope the study will benefit the long suffering patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnosis of PD41 or MSA43 based on the established consensus criteria
2. Age above 30 years old and below 85 years

Exclusion Criteria:

1. Impairment of cognition that leads unable to fully cooperate with the oral commands during examinations
2. Functional III or above congestive heart failure, or cancer with distant metastasis
3. Hoehn and Yahr stage 5 in PD or MSA

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
EEG recording before and after the tDCS session | baseline to week 4
  Gait recording by 64 channels EEG device. Four different frequency bands ( theta, alpha, beta, and gamma) will be investigated. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.

SECONDARY OUTCOMES:
Electromyography recording before and after the tDCS session | baseline to week 4
  The 4 pairs of leg EMG recording during 50 meters walking. The EMG signals will be filtered with a band pass ranging from 0.05 to 70 Hz. Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III before and after the tDCS session | baseline to week 4
  UPDRS contains four parts, the third part of which is reported in this outcome. Part III is clinician-scored monitored motor evaluation (14 questions, ranges from 0=normal to 4= Severe). The scoring of Part III varies between 0-56. The higher score indicates the worse motor function. Negative change from baseline values indicate improvement.
Change in Unified Multiple System Atrophy Rating Scale (UMSARS) subscores (UMSARS-1 and UMSARS-2) before and after the tDCS session | baseline to week 4
  UMSARS contains four parts, the UMSARS-1 and UMSARS-2 are reported in this outcome. UMSARS-1 scores symptoms of neurological and autonomic dysfunction (12 questions). UMSARS-2 is motor examination (14 questions). All questions range from 0 (normal) to 4(extreme dysfunction). Higher scores mean greater the impairment. Negative change from baseline values indicate improvement.

OTHER OUTCOMES:
Change in New freezing of gait questionnaire (NFOG-Q) before and after the tDCS session | baseline to week 4
  NFOG-Q contains three parts: in the first part, a video clip will be shown to the participants with PD and help to classify whether an individual is a freezer or non-freezer. The second and third part of the questionnaire is designed for freezers only. Par II (items 2-6, scores range between 0-19) assesses the severity of FOG according to the frequency and duration of the freezing episodes. Part III (items 7-9, scores range between 0-9) evaluates the impact of freezing on daily activities. The higher score indicates the worse freezing of gait. Negative change from baseline values indicate improvement.
Change in Tinetti's Mobility Index total score before and after the tDCS session | baseline to week 4
  The Tinetti's Mobility Index contains two parts, Part I is Balance tests (9 questions, scores range between 0-16) and Part II is Gait tests (7 questions, scores range between 0-12). The scoring of this scale varies between 0 and 28 (< 19 high fall risk, 19-24 medium fall risk, 25-28 low fall risk). Negative change from baseline values indicate increased fall risk.
Change inParkinson's Disease Questionnaire 39 (PDQ-39) before and after the tDCS session | baseline to week 4
  PDQ-39 is composed of 39 questions, divided into 8 parts: mobility, activities of daily living (ADLs), emotional well-being, stigma, social support, cognition, communication and physical discomfort. It assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living. All questions range from 0 to 4 (0=never, 4=always). The scoring of this scale varies between 0-156. Negative change from baseline values indicate better quality of life rating.
Change in Short Form 36 Health Survey (SF-36) total score before and after the tDCS session | baseline to week 4
  SF-36 is composed of 36 questions, divided into 8 parts: Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health. The scores are weighted sums of the questions in each section. Scores range from 0-100 (Lower scores = more disability, higher scores = less disability). Negative change from baseline values indicate worse quality of life rating.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan